CLINICAL TRIAL: NCT00673504
Title: Prospective Randomized Phase II Trial With Gemcitabine Plus Sunitinib Versus Gemcitabine Alone in First-line Therapy of Metastatic or Locally Advanced Pancreatic Cancer
Brief Title: First-Line Gemcitabine Chemotherapy With Our Without Sunitinib In Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central European Society for Anticancer Drug Research (Other)
Responsible Party: Central European Society for Anticancer Drug Research-EWIV, Non-Profit Otrganization Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-II-004 / 2007-005022-71
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Pancreatic Cancer
Keywords: cancer; pancreatic cancer; gemcitabine; sunitinib; Phase 2
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Gemcitabine; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Gemcitabine + Sunitinib
  Interventions: Drug: Gemcitabine + Sunitinib
- B (Other): Gemcitabine
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine + Sunitinib — Gemcitabine 1.000 mg/m2, d1,8q3weeks Sunitinib 50 mg/day (2weeks on/1weeks off)
  Arms: A
Drug: Gemcitabine — 1.000 mg/m2 d1,8,15q4weeks
  Arms: B

SUMMARY:
Primary objective: to evaluate whether the addition of sunitinib prolongates the Progression-Free Survival (PFS) in patients with advanced pancreatic cancer receiving first-line gemcitabine chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffer from locally advanced or metastatic pancreatic cancer
* Patients with measurable disease (at least one uni-dimensionally measurable target lesion by CT-scan or MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST).
* ECOG performance status 0 to 1
* Signed written informed consent.
* White blood cell count (WBC) >= 3x10^9/L with neutrophils >= 1.5 x 10^9/L, platelet count >= 100x10^9/L, hemoglobin >= 5.6 mmol/L (9 g/dL).
* Total bilirubin < 2 x upper limit of normal.
* AST and ALT < 2.5 x upper limit of normal, or < 5 x upper limit of normal in case of liver metastases.
* Serum creatinine < 1.5 x upper limit of normal
* Normal ECG without QT prolongation

Exclusion Criteria:

* Resectable pancreatic cancer
* Previous chemotherapy (for adjuvant or metastatic disease)
* Any investigational drug within the 30 days before inclusion.
* Prior use of sunitinib or other multitarget tyrosine kinase inhibitor
* Pregnancy (absence to be confirmed by beta-hCG test) or lactation period.
* Men or women of child-bearing potential who are sexually active and unwilling to use a medically acceptable method of contraception during the trial.
* Clinically symptomatic brain or meningeal metastasis. (known or suspected)
* Cardiac arrhythmias requiring anti-arrhythmics (excluding beta blockers or digoxin).
* History of any of the following cardiac events within the past 6 months: myocardial infarction (including severe/unstable angina; coronary/peripheral artery bypass graft; symptomatic congestive heart failure (CHF) > NYHA Class II; cerebrovascular accident or transient ischemic attack; pulmonary embolism
* Uncontrolled severe hypertension (failure of diastolic blood pressure to fall below 90 mm Hg despite the use of up to 3 anti-hypertensive drugs
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease or chronic diarrhea
* Previous malignancy (other than pancreatic cancer) in the last 5 years except basal cell cancer of the skin, pre-invasive cancer of the cervix or superficial bladder tumor [Ta, Tis and T1].
* History of organ allograft
* Patients requiring long-term cortisone therapy
* Patients requiring oral anticoagulation treatment (such as marcoumar)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-04; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Time to Progression | once all patients completed treatment

SECONDARY OUTCOMES:
Response Rate (RR) | once all patients completed treatment
overall survival | at study end
Safety | at study end

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (10):
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Universitätsklinikum Essen, Essen
  - Krankenhaus, Frankfurt
  - Klinikum der J. W. Goethe Universität; Zentrum der Inneren Medizin, Frankfurt
  - Internistisches Facharztzentrum, Frankfurt
  - Martin-Luther-Universität Halle-Wittenberg; Medizinische Fakultät, Halle
  - Facharztpraxis, Heidelberg
  - Klinikum Lüdenscheid, Lüdenscheid
  - Klinikum Nürnberg Nord, Nuremberg
  - Robert-Bosch-Krankenhaus, Stuttgart
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- See also: German Study Description on CESAR's homepage — http://www.cesar.or.at/main.asp?VID=1&kat1=49&kat2=370&kat3=&Text=&SSSID=5